CLINICAL TRIAL: NCT01960036
Title: Body-oriented Therapy for Womens Substance Use Disorder Treatment
Brief Title: Body-oriented Therapy for Women in SUD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Cynthia Price, Research Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 46102-J; R01DA033324 (NIH)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Substance Use Disorder
Keywords: Substance Use Disorders; Complementary Therapies; Women; Mind-Body Therapies; Behavior and Behavior Mechanisms
MeSH Terms: conditions — Substance-Related Disorders; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment as usual (TAU) (No Intervention): Usual intensive outpatient treatment for substance use disorders
- Mindful Awareness in Body-oriented Therapy (MABT) (Experimental): A mind-body intervention to teach interoceptive skills for self-care.
  Interventions: Behavioral: Mindful Awareness in Body-oriented Therapy
- Womens Health Education (Active Comparator): A comparative arm to control for time and attention that involves education about the human body relevant to women's health.
  Interventions: Behavioral: Womens Health Education

INTERVENTIONS:
Behavioral: Mindful Awareness in Body-oriented Therapy
  Arms: Mindful Awareness in Body-oriented Therapy (MABT)
Behavioral: Womens Health Education
  Arms: Womens Health Education

SUMMARY:
The long-term objective of this study is to improve women's substance use disorder (SUD) treatment. The immediate project goal is to test the efficacy of an innovative mind-body intervention, Mindful Awareness in Body-Oriented Therapy (MABT) to reduce substance use relapse among women in SUD treatment.

A novel mind-body approach, MABT combines a hands-on (manual) approach with mind-body psycho-education approaches of interoceptive training and mindfulness to develop somatically-based self-care skills and to facilitate emotion regulation. A three-group, randomized clinical trial using repeated measures, this project will enroll and randomize 225 women to one of three groups, MABT + Treatment-as-usual (TAU) (n=75), TAU only (n=75), and Women's Health Education (WHE) + TAU (to control for time and attention) (n=75). Study conditions will be compared at baseline, post-intervention, and at 6 and 12 month follow-up.

The primary aim is to test the hypothesis that MABT will result in reduced substance use and related health outcomes compared to TAU and to WHE+ TAU at 12 month follow-up. The second aim is to examine hypothesized underlying mechanisms of MABT. Female outpatients in two diverse community treatment facilities, serving racially diverse patients, will be recruited for study participation. This study builds on promising preliminary evidence of MABT feasibility and acceptability in substance use disorder treatment for women, and addresses the need for more clinical research aimed at improving SUD treatment outcomes for women.

ELIGIBILITY:
Inclusion Criteria:

* 1) female, 2) enrolled in intensive outpatient (IOP) with at least 8 weeks remaining in planned SUD treatment program, 3) agrees to forgo (non-study) manual therapies (e.g.,massage) and mind-body therapies (e.g., mindfulness meditation) for 3 months (baseline to post-test); 4) willing to sign release for access of electronic medical records; 5) fluent in English; and 6) can attend MABT and WHE sessions when offered.

Exclusion Criteria:

* ) untreated psychotic diagnosis or symptoms, using modules from the MINI International Neuropsychiatric Interview; 2) unwilling or unable to remain in treatment for the duration of the trial (includes planned relocation, pending incarceration, planned surgical procedures, etc.); 3) cognitive impairment, to be assessed with an informed consent quiz, followed by the Mini-Mental Status Exam (MMSE), a common screening tool in SUD treatment studies, if there is demonstrated difficulty comprehending the consent; or 4) currently pregnant.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Timeline Follow-back Interview (TLFB) | Change from baseline in TLFB assessed at different time points (3,6 and 12 months)
  Collects self-report substance use information using a calendar method

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Price, PhD, MA, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Price CJ, Wells EA, Donovan DM, Rue T. Mindful awareness in body-oriented therapy as an adjunct to women's substance use disorder treatment: a pilot feasibility study. J Subst Abuse Treat. 2012 Jul;43(1):94-107. doi: 10.1016/j.jsat.2011.09.016. Epub 2011 Nov 25. PMID 22119181
- [Background] Price CJ, Wells EA, Donovan DM, Brooks M. Implementation and acceptability of Mindful Awareness in Body-oriented Therapy in women's substance use disorder treatment. J Altern Complement Med. 2012 May;18(5):454-62. doi: 10.1089/acm.2011.0126. Epub 2012 Apr 23. PMID 22524991
- [Background] Price CJ, Crowell SE. Respiratory sinus arrhythmia as a potential measure in substance use treatment--outcome studies. Addiction. 2016 Apr;111(4):615-25. doi: 10.1111/add.13232. Epub 2016 Jan 5. PMID 26567088